CLINICAL TRIAL: NCT02237209
Title: A Phase I Study of the Safety and Immunogenicity of Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine RSV LID ΔM2-2 in RSV-Seronegative Infants and Children
Brief Title: Safety and Immune Response to a Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccine in RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2000; DAIDS ES (Registry Identifier: 12016)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSV LID ΔM2-2 Vaccine (Experimental): Participants will receive one dose of the RSV LID ΔM2-2 vaccine at study entry, delivered as nose drops.
  Interventions: Biological: RSV LID ΔM2-2 Vaccine
- Placebo Vaccine (Placebo Comparator): Participants will receive one dose of placebo at study entry, delivered as nose drops.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: RSV LID ΔM2-2 Vaccine — 10^5.0 plaque forming units (PFU); 0.5 mL dose delivered as nose drops (approximately 0.25 mL per nostril)
  Arms: RSV LID ΔM2-2 Vaccine
Biological: Placebo Vaccine — 0.5 mL dose delivered as nose drops (approximately 0.25 mL per nostril)
  Arms: Placebo Vaccine

SUMMARY:
Respiratory syncytial virus (RSV) is a common cause of illness in infants and children around the world. This study will evaluate the safety and immune response to an RSV vaccine in RSV-seronegative infants and children.

This study is a companion study to CIR 291.

DETAILED DESCRIPTION:
RSV is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age in the world. RSV illness can range from mild upper respiratory tract illness (URI) to severe LRI, including bronchiolitis and pneumonia. Severe RSV disease in infancy may also predispose children to develop reactive airway disease during childhood. The purpose of this study is to evaluate the safety and immunogenicity of an RSV vaccine (RSV LID ΔM2-2) in RSV-seronegative infants and children at least 6 months and through 24 months of age.

To determine study eligibility, the screening process will include a blood collection. Screening may begin after the RSV season (i.e., as of April 1) and enrollment must precede the RSV season (no later than October 14). At study entry, eligible participants will be randomly assigned to receive one dose of either the RSV vaccine or placebo, which will be delivered as nose drops. Participants will also undergo a review of medical history, clinical assessment, and a nasal wash. They will then receive their assigned vaccine and will remain under observation for monitoring for 30 minutes after receiving the vaccine. Additional study visits will occur at Days 3, 5, 7, 10, 12, 14, 17, 19, 21, 28, and 56. These visits will include clinical assessments and nasal washes; on Day 56, a blood collection will also occur. On days where no study visit is scheduled (through Day 29), participants' parents or guardians will report participants' temperatures and signs of illness to researchers by e-mail or phone.

In October following vaccination, participants may have a pre-RSV season blood collection visit. During RSV season, November through March following vaccination, researchers will contact participants' parents or guardians on a weekly basis for follow-up monitoring. During this time frame, participants seen by a medical provider for fever, respiratory illness, or otitis media will have a study visit, which will include a nasal wash and clinical assessment. In April following vaccination, participants will undergo a final blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 6 months (defined as at least 180 days) of age at the time of screening and less than 25 months (defined as less than 750 days) of age
* Participant is in good health based on review of the medical record, history, and physical examination, without evidence of chronic disease. Note: any questions regarding interpretation of this criterion should be forwarded to the team.
* Parents/guardians demonstrate their understanding of the study, sign the informed consent, and agree to administration of study product following a detailed explanation of the study
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening obtained no more than 42 days prior to scheduled inoculation
* Has a current height and weight above the 5th percentile for age
* Participant has received routine immunizations appropriate for age. Prior vaccines were administered at least:

  * 2 weeks prior to enrollment for inactivated and subunit vaccines and rotavirus vaccine, and
  * 4 weeks prior to enrollment for all other live vaccines.
* Participant is expected to be available for the duration of the study
* If born to an HIV-infected woman, participant must be non-breastfeeding with documentation of two negative HIV nucleic acid (RNA or DNA) tests with both collected when at least 1 month of age and at least one collected when at least 4 months of age, and no positive HIV nucleic acid (RNA or DNA) test; or two negative HIV antibody tests, both collected at less than or equal to 6 months of age

Exclusion Criteria:

* Known or suspected HIV infection or impairment of immunological functions
* Receipt of immunosuppressive therapy, including any systemic corticosteroids within 30 days of enrollment. Note: Cutaneous (topical) steroid treatment is not an exclusion.
* Bone marrow/solid organ transplant recipient
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities
* Previous receipt of a licensed or investigational RSV vaccine (or placebo) or previous receipt of or planned administration of any anti-RSV product (such as ribavirin or RSV IG)
* Previous vaccine-associated anaphylactic or other severe adverse vaccine reaction
* Known hypersensitivity to any study product component
* Heart disease. Note: Participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment may be enrolled.
* Lung disease, including any history of wheezing or reactive airway disease
* Member of a household that contains, or will contain, an infant who is less than 6 months of age at the enrollment date through Day 28
* Member of a household that contains another child who is, or is scheduled to be, enrolled in IMPAACT 2000, and there has been or will be an overlap in residency during that other child's participation in the study's Acute Phase (Days 0 to 28)
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is greater than or equal to 5 years of age with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell count less than 300/mcL. CD4 T lymphocyte count must have been measured within 6 months prior to enrollment; or
  * a person less than 5 years of age with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 15. CD4 T lymphocyte percentage must have been measured within the 6 months prior to enrollment; or
  * a person who has received chemotherapy within the 12 months prior to enrollment.
  * Verbal report of CD4 T cell lymphocyte is sufficient documentation if the parent/guardian is confident of history.
* Attends a daycare facility and shares a room with infants less than 6 months of age, and parent/guardian is unable or unwilling to suspend daycare for 28 days following inoculation.
* Any of the following events at the time of enrollment:

  * fever (rectal temperature of greater than or equal to 100.4°F [38°C]), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis), or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media.
* Receipt of the following prior to enrollment:

  * any killed vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior.
* Scheduled administration of the following after planned inoculation:

  * killed vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or drug in the 28 days after.
* Receipt of immunoglobulin, any antibody products, or any blood products
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, antiparasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below. Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Receipt of salicylate (aspirin) or salicylate-containing products within the past month
* Born at less than 37 weeks gestation and less than 1 year of age at the time of enrollment
* Meets criteria for failure to thrive within the 6 months prior to enrollment: a decline in height or weight growth that has crossed two major growth percentiles (e.g., from above the 75th to below the 25th) in an interval of less than 6 months
* Suspected or documented developmental disorder, delay, or other developmental problem

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related solicited adverse events (AEs) that occur during the acute monitoring phase of the study, the first 28 days after inoculation | Measured through Day 28
Severity of vaccine-related solicited AEs that occur during the acute monitoring phase of the study, the first 28 days after inoculation | Measured through Day 28
Frequency of vaccine-related lower respiratory illness | Measured through Day 56
Proportion of participants that develop 4-fold or greater rises in RSV-neutralizing antibody titer following vaccination | Measured through Day 56
  Antibody responses to the RSV F glycoprotein will also be assessed by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McFarland, MD, Study Chair — Children's Hospital Colorado
Locations (7):
- United States (7):
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Johns Hopkins University Center for Immunization Research, Baltimore, Maryland
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee

REFERENCES:
- [Derived] McFarland EJ, Karron RA, Muresan P, Cunningham CK, Valentine ME, Perlowski C, Thumar B, Gnanashanmugam D, Siberry GK, Schappell E, Barr E, Rexroad V, Yogev R, Spector SA, Aziz M, Patel N, Cielo M, Luongo C, Collins PL, Buchholz UJ; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) 2000 Study Team. Live-Attenuated Respiratory Syncytial Virus Vaccine Candidate With Deletion of RNA Synthesis Regulatory Protein M2-2 is Highly Immunogenic in Children. J Infect Dis. 2018 Apr 11;217(9):1347-1355. doi: 10.1093/infdis/jiy040. PMID 29509911